CLINICAL TRIAL: NCT00725231
Title: Phase III Study of CHOP-14 Plus or Minus Alemtuzumab in Peripheral T-cell Lymphoma of the Elderly
Brief Title: Immunotherapy in Peripheral T Cell Lymphoma - the Role of Alemtuzumab in Addition to Dose Dense CHOP
Acronym: A-CHOP-14
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Göttingen (Other)
Collaborators: German High-Grade Non-Hodgkin's Lymphoma Study Group (Other); Nordic Lymphoma Group (Network)
Responsible Party: Principal Investigator, Prof. Dr. Lorenz Trümper, Head of Departement of Haemtology and Oncology, University of Göttingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSHNHL 2006-1B / ACT-2; BMBF GFVT 01014715
Record Dates: First submitted 2008-07-25; First posted 2008-07-30 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Peripheral T Cell Lymphoma, Unspecified; Angioimmunoblastic Lymphadenopathy; Extranodal NK/T-cell Lymphoma
Keywords: T cell lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Extranodal NK-T-Cell | interventions — Alemtuzumab; Drug Therapy; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Chemotherapy with dose dense CHOP-14, 6 cycles
  Interventions: Drug: chemotherapy
- Arm B (Experimental): Chemotherapy with dose dense CHOP-14, 6-cycles, together with 30mg Alemtuzumab s.c. for the first 4 cycles
  Interventions: Biological: alemtuzumab; Drug: chemotherapy

INTERVENTIONS:
Biological: alemtuzumab — Addition of 30 mg Alemtuzumab by subcutaneous application for the first 4 cycles
  Other Names: monoclonal anti CD52 antibody
  Arms: Arm B
Drug: chemotherapy — dose dense chemotherapy with CHOP-14, 6 cycles, + G-CSF
  Other Names: chemotherapy cylcophosphamide, hydroxyldaunorubicin

SUMMARY:
Peripheral T cell lymphomas comprise 10-15% of all malignant lymphomas. The prognosis is significantly worse than that of aggressive B cell lymphomas. The prospects of elderly patients are especially poor, with an estimated disease free survival of only 25% after three years. Previous phase II trials have demonstrated a significant activity of the monoclonal anti CD52 antibody alemtuzumab in primary and relapsed T cell lymphoma. The investigators thus propose to investigate the value of adjuvant alemtuzumab in combination with dose dense CHOP-14 in patients with previously untreated peripheral T cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* all risk groups of peripheral T cell lymphoma
* performance status ECOG 0-2
* written consent
* measurable disease

Exclusion Criteria:

* stage I N without bulky disease
* already initiated treatment
* serious accompanying disorder or impaired organ function
* bone marrow involvement >25%
* HIV positivity
* leukemic manifestation of lymphoma
* simultaneous participation in another trial
* platelets < 100 000/ mm, leukocytes < 2500 /mm

Ages: 61 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2008-02; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 3 years

SECONDARY OUTCOMES:
Rate of complete and partial remissions | 4 months after inclusion
treatment related deaths | time of occurence
Overall survival | @ 3 years
protocol adherence | 4 months of treatment
immune reconstitution after alemtuzumab CHOP | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz H Trümper, MD, Principal Investigator — University of Göttingen
Locations (1):
- University of Göttingen, Göttingen, Lower Saxony, Germany